CLINICAL TRIAL: NCT04906772
Title: Dexmedetomidine-ketamine Versus Propofol-ketamine for Sedation During Upper Gastro-intestinal Endoscopy in Hepatic Patients (a Comparative Randomized Study)
Brief Title: Dexmedetomidine-ketamine Versus Propofol-ketamine for Sedation During Endoscopy in Hepatic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tamer Nabil Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Tamer Nabil Abdelrahman, lecturer of anaesthesia, intensive care and pain management, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAMSU R 21
Record Dates: First submitted 2021-02-27; First posted 2021-05-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia; Reaction
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group KD (Experimental): participants received loading of ketamine 1 mg/kg and dexmedetomidine 1µg/kg over 10 minutes then continue by a dose of 0.25 mg/kg/hr ketamine and 0.25µg/kg/hr dexmedetomidine throughout the procedure.
  Interventions: Drug: Dexmedetomidine
- Group KP (Active Comparator): participants received loading of ketamine 1 mg/kg and propofol 1 mg/kg over 10 minutes then continue by a dose of 0.25 mg/kg/hr propofol and 0.25 µg/kg/hr dexmedetomidine throughout the procedure.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — participants received loading of ketamine 1 mg/kg and dexmedetomidine 1µg/kg over 10 minutes then continue by a dose of 0.25 mg/kg/hr ketamine and 0.25µg/kg/hr dexmedetomidine throughout the procedure.
  Other Names: ketamine
  Arms: Group KD
Drug: Propofol — participants received loading of ketamine 1 mg/kg and propofol 1mg/kg over 10 minutes then continue by a dose of 0.25 mg/kg/hr propofol and 0.25µg/kg/hr dexmedetomidine throughout the procedure.
  Other Names: ketamine
  Arms: Group KP

SUMMARY:
We aim to compare the response to ketamine/dexmedetomidine and ketamine/propofol combinations used in hepatic patients with child-Pugh classification (class A), and early (class B) undergoing UGIE.

DETAILED DESCRIPTION:
70 Patients will be randomly allocated into two groups; Group (KD): Ketamine/dexmedetomidine (35 patients), will receive IV ketamine 0.25mg/kg and dexmedetomidine1µg/kg over 10 min as loading followed by dexmedetomidine infusion with a rate of 0.5µg/kg/hr and Group (KP): ketamine/propofol (35 patients) will receive IV ketamine 0.25 mg/kg loading and propofol 1 mg/kg over 10 min followed by propofol infusion with a rate of 0.5 mg/kg/hr as a control group.

ELIGIBILITY:
Inclusion Criteria:

* hepatic patients with child-Pugh classification (class A), and (class B)
* American Society of Anesthesiologists physical status II, III
* aged 18 to 60 years
* scheduled for elective Upper gastro-intestinal endoscopy.

Exclusion Criteria:

* emergency gastro-intestinal endoscopy.
* patients with severe hepatic disorder (Child C) ,
* chronic neuro-psychiatric disorder,
* history of neuro-psychiatric drug intake,
* severe cardiovascular diseases,
* pregnancy,
* history of drug abuse, and
* history of allergy to any of the used drugs in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
induction time | after 5 minutes from the start of drug infusion till target Ramsay Sedation Score ≥ 3 is reached
  Time to reach target Ramsay Sedation Score ≥ 3
Recovery time | after 10 minutes from the stoppage of drug infusion at the end of the procedure till spontaneous eye opening
  time from the stoppage of drug infusion at the end of the procedure till spontaneous eye opening

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain-Shams university, Cairo, Egypt